CLINICAL TRIAL: NCT05299151
Title: The Effect of Vestibular Rehabilitation on the Kinetic and Kinematic Parameters of Walking in Patients With Multiple Sclerosis
Brief Title: Gait Analysis in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Kültür University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Ertürk, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: VR-1
Record Dates: First submitted 2022-03-09; First posted 2022-03-28 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis; 3D Gait Analysis; Vestibular Rehabilitation
Keywords: gait analysis, multiple sclerosis, vestibular, kinetic, kinematic
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation Group (Experimental): A vestibular rehabilitation exercise program, which is determined based on the literature and personalized according to the functional disabilities of each patient, will be applied to the participants in the experimental group. An exercise session will be performed for a total of 40 minutes, with each exercise for 1-2 minutes. Exercise training will be applied 2 days a week for 8 weeks and they will be asked to do it at home once a week.
  Interventions: Other: Vestibular exercises
- Standard Neurorehabilitation Group (Active Comparator): A neurorehabilitation program based on stretching, strengthening, posture, mobilization, static and dynamic balance exercises will be applied. Each training session will be 40 minutes in total. Exercise training will be done in the clinical setting 2 days a week for 8 weeks, and they will be asked to do it at home once a week.
  Interventions: Other: Standard neurorehabilitation exercises

INTERVENTIONS:
Other: Vestibular exercises — The vestibular exercise program basically consists of 3 groups of exercises: adaptation, substitution, and habituation exercises. It is aimed to provide vestibular adaptation with adaptation exercises. Exercises that include visual and somatosensory cues to improve gaze and postural stability constitute substitution exercises. Balance exercises can be performed with eyes open and closed, or somatosensory cues can be changed by performing them on soft ground. Removing or reducing clues allows the patient to use other systems as well. The basis of habituation exercises is the reduction of the pathological response as a result of repeated exposure to the provocative stimulus. Habituation is specific to the type, intensity, and direction of stimuli. In most cases, the movement that stimulates the pathological response is less frequently performed during daily activities and promotes compensation for the initially abnormal signal of treatment.
  Arms: Vestibular Rehabilitation Group
Other: Standard neurorehabilitation exercises — A neurorehabilitation program based on stretching, strengthening, posture, mobilization, static and dynamic balance exercises (standing on one leg, tandem, balance board, etc.) will be applied.
  Arms: Standard Neurorehabilitation Group

SUMMARY:
In the literature, the results of vestibular rehabilitation treatment applied in patients with Multiple Sclerosis (MS) have been investigated in detail under the headings such as fatigue, physical activity level, and quality of life, and its effects on walking have also been tried to be examined. However, in the studies conducted, gait assessments were made through questionnaires and timed tests, and devices that provide more objective data such as 3-dimensional gait analysis were not used. Again, the effects of vestibular rehabilitation programs on dual-task were not examined in previous studies.

Therefore, the aims of our study are:

1. To determine the effect of individually designed vestibular rehabilitation exercises on the kinetic and kinematic components of walking;
2. To determine the effect of vestibular rehabilitation exercises specially designed for the person on gait parameters during cognitive and motor tasks.

ELIGIBILITY:
Inclusion Criteria:

* Between aged 25-60 years
* Diagnosed with MS for at least 5 years
* Relapsing and progressive MS according to Mc Donald criteria
* EDSS score of ≤ 3.5 ≤ 6
* Modified Ashworth Scale < 3
* Being eligible to work by a neurologist

Exclusion Criteria:

* Having had an MS-related attack in the 3 months before the study
* Changes in medications within 6 months prior to the study
* To have participated in the rehabilitation program within 1 month before the study
* Serious neurological, cardiac, pulmonary, rheumatological, audiovisual, or orthopedic disorders that limit assessments and/or intervention programs

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
3D Gait Analysis System - pre assesment | It will be done at the beginning of the study. An analysis session lasts nearly 2 hours per patient. Evaluation of all participants will take approximately 2 months.
  Kinetic and kinematic data of gait will be collected in the motion analysis laboratory using 6 infrared digital cameras (Vantage 5.0), 2 synchronized video cameras (Vicon Vue) and 2 force platforms (AMTI).
3D Gait Analysis System - post assesment | It will be done at the end of the study. An analysis session lasting nearly 2 hours per patient. Evaluation of all participants will take approximately 2 months.
  Kinetic and kinematic data of gait will be collected in the motion analysis laboratory using

SECONDARY OUTCOMES:
One Leg Standing Test - pre assesment | It will be done at the beginning of the study. The test lasts nearly 5 minutes.
  It will be used to determine the patient's standing balance. The duration of standing on one leg will be recorded with a stopwatch and 3 repetitions will be taken and the most successful score will be used in the analysis.
One Leg Standing Test - post assessment | It will be done at the end of the study. The test lasts nearly 5 minutes.
  It will be used to determine the patient's standing balance. The duration of standing on one leg will be recorded with a stopwatch and 3 repetitions will be taken and the most successful score will be used in the analysis.
Dizziness Handicap Inventory - pre assessment | It will be done at the beginning of the study. The test lasts nearly 15 minutes.
  The Dizziness Disability Inventory consists of 25 items that determine the aggravating factors of patients' dizziness and balance disorder, as well as emotional and functional outcomes in vestibular system diseases. It includes 9 items that determine emotional and functional status, and seven items that determine physical function.
Dizziness Handicap Inventory - post assessment | It will be done at the end of the study. The test lasts nearly 15 minutes.
  The Dizziness Disability Inventory consists of 25 items that determine the aggravating factors of patients' dizziness and balance disorder, as well as emotional and functional outcomes in vestibular system diseases. It includes 9 items that determine emotional and functional status, and seven items that determine physical function.
2 Minute Walking Test - pre assessment | It will be done at the beginning of the study. The test lasts nearly 5 minutes.
  The distance that patients will walk for 2 minutes will be measured and recorded.
2 Minute Walking Test - post assessment | It will be done at the end of the study. The test lasts nearly 5 minutes.
  The distance that patients will walk for 2 minutes will be measured and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpaşa, Vocational School of Health Services, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Comber L, Galvin R, Coote S. Gait deficits in people with multiple sclerosis: A systematic review and meta-analysis. Gait Posture. 2017 Jan;51:25-35. doi: 10.1016/j.gaitpost.2016.09.026. Epub 2016 Sep 26. PMID 27693958
- [Background] Huisinga JM, Schmid KK, Filipi ML, Stergiou N. Gait mechanics are different between healthy controls and patients with multiple sclerosis. J Appl Biomech. 2013 Jun;29(3):303-11. doi: 10.1123/jab.29.3.303. Epub 2012 Aug 22. PMID 22923390
- [Background] Garcia-Munoz C, Cortes-Vega MD, Heredia-Rizo AM, Martin-Valero R, Garcia-Bernal MI, Casuso-Holgado MJ. Effectiveness of Vestibular Training for Balance and Dizziness Rehabilitation in People with Multiple Sclerosis: A Systematic Review and Meta-Analysis. J Clin Med. 2020 Feb 21;9(2):590. doi: 10.3390/jcm9020590. PMID 32098162
- [Background] Gunn H, Markevics S, Haas B, Marsden J, Freeman J. Systematic Review: The Effectiveness of Interventions to Reduce Falls and Improve Balance in Adults With Multiple Sclerosis. Arch Phys Med Rehabil. 2015 Oct;96(10):1898-912. doi: 10.1016/j.apmr.2015.05.018. Epub 2015 Jun 10. PMID 26070975